CLINICAL TRIAL: NCT03533894
Title: French Observational Study With Colic Capsule
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: ONECC
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Colic Capsule Interest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: colic capsule — colic polyp diagnosis

SUMMARY:
colic capsule usings with patients without possible colic endoscopy

ELIGIBILITY:
Inclusion Criteria:

* anesthesia not possible
* incomplete colic endoscopy
* colic endoscopy refused

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: men or women with colic endoscopy problems
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
number of polyps or lesions | 5 years
  number of polyps or lesions

IPD SHARING:
Plan to Share IPD: Undecided